CLINICAL TRIAL: NCT01977703
Title: Prospective Randomized Evaluation of an Ultra Conservative Approach to Implantable Defibrillator (ICD) Programming in Patients With a Left Ventricular Assist Device (LVAD).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Principal Investigator, Christopher Ellis, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 131336
Record Dates: First submitted 2013-10-30; First posted 2013-11-07 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Heart Failure
Keywords: Heart Failure; Advanced Heart Failure; LVAD; Left Ventricular Assist Device; Heart-Assist Devices
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional ICD Programming (Active Comparator): ICD will be set to pre-LVAD settings post LVAD implant.
  Interventions: Other: Traditional ICD Programming
- Ultra Conservative ICD Programming (Experimental): ICD will be set to ultra conservative settings post LVAD implant.
  Interventions: Other: Ultra Conservative ICD Programming

INTERVENTIONS:
Other: Ultra Conservative ICD Programming
  Arms: Ultra Conservative ICD Programming
Other: Traditional ICD Programming
  Arms: Traditional ICD Programming

SUMMARY:
We propose to study a strategy empirically applied for the past 6 months at a high volume LVAD center (Vanderbilt Heart and Vascular Institute). This utilizes an ultra conservative device programming strategy to maximize battery longevity, avoid inappropriate implantable cardioverter defibrillator (ICD) therapy, improve quality of life through reduction in overall shock burden, and potentially avoid unnecessary device generator changes prior to transplant. Avoiding CIED (cardiac implantable electronic device) change out device procedures prior to transplant is desirable.

ELIGIBILITY:
Inclusion:

* Age ≥ 18
* Advanced Heart Failure
* Scheduled for Heartmate II LVAD implant
* With existing ICD

Exclusion:

-Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Time to first ICD shock following LVAD implant | Within 12 months following LVAD implant

SECONDARY OUTCOMES:
Frequency of anti-tachycardia pacing (ATP) therapy administration for appropriate or inappropriate arrhythmia detection | Within 12 months following LVAD implant
  Number of ATP occurrences
Frequency of ICD generator change prior to definitive therapy | Within 12 months following LVAD implant
  Number of patients requiring ICD generator change
Cardiac implantable electronic device (CIED) battery voltage/estimated longevity changes | Within 12 months following LVAD implant
  Battery voltage and battery life measured in days
Frequency of arrhythmic syncope | Within 12 months following LVAD implant
  Number of syncope occurrences
Hospitalization frequency for decompensated congestive heart failure | Within 12 months following LVAD implant
  Number of hospitalizations
Determine survival to heart transplantation following LVAD implant | Within 12 months following LVAD implant
  Number of patients, post LVAD implant, to receive heart transplant and number of survival days post implant

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ellis, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Richardson TD, Hale L, Arteaga C, Xu M, Keebler M, Schlendorf K, Danter M, Shah A, Lindenfeld J, Ellis CR. Prospective Randomized Evaluation of Implantable Cardioverter-Defibrillator Programming in Patients With a Left Ventricular Assist Device. J Am Heart Assoc. 2018 Feb 23;7(5):e007748. doi: 10.1161/JAHA.117.007748. PMID 29475875